CLINICAL TRIAL: NCT04996771
Title: A Phase Ⅰb/II Study of Surufatinib Combined With Chemotherapy Plus Toripalimab or Not in Patients With Small Cell Lung Cancer
Brief Title: Surufatinib Combined With Chemotherapy Plus Toripalimab or Not in the Treatment of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-L103
Record Dates: First submitted 2021-08-05; First posted 2021-08-09 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — surufatinib; PE regimen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib Combined With Toripalimab and Chemotherapy (Experimental)
  Interventions: Drug: Surufatinib,Etoposide,Cisplatin,Toripalimab
- Surufatinib Combined With Chemotherapy (Experimental)
  Interventions: Drug: Surufatinib,Etoposide,Cisplatin

INTERVENTIONS:
Drug: Surufatinib,Etoposide,Cisplatin,Toripalimab — In dose escalation, Surufatinib and will be administered orally (PO) once daily (QD) ,d1-21，q3w+Toripalimab 240mg,d1,q3w+Etoposide 100mg/m2,d1-3,q3w+Cisplatin 75mg/m2 , d1, q3w,4 cycles in total.
  At the indication-specific expansion portion of the study, patients will receive surufatinib RP2D,d1-21，q3w+Toripalimab 240mg,d1,q3w+Etoposide 100mg/m2,d1-3,q3w+Cisplatin 75mg/m2 , d1, q3w,4 cycles in total. After the end of the first-line treatment, patients with CR, PR, and SD can continue to maintenance treatment with Surufatinib RP2D,d1-21，q3w＋Toripalimab 240mg,d1,q3w was taken orally until the disease progressed.
  Arms: Surufatinib Combined With Toripalimab and Chemotherapy
Drug: Surufatinib,Etoposide,Cisplatin — In dose escalation, Surufatinib and will be administered orally (PO) once daily (QD) ,d1-21，q3w+Etoposide 100mg/m2,d1-3,q3w+Cisplatin 75mg/m2 , d1, q3w,4 cycles in total.
  At the indication-specific expansion portion of the study, patients will receive surufatinib RP2D,d1-21，q3w+Etoposide 100mg/m2,d1-3,q3w+Cisplatin 75mg/m2 , d1, q3w,4 cycles in total. After the end of the first-line treatment, patients with CR, PR, and SD can continue to maintenance treatment with Surufatinib RP2D,d1-21，q3w was taken orally until the disease progressed.
  Arms: Surufatinib Combined With Chemotherapy

SUMMARY:
To evaluates the effectiveness and safety of Surufatinib combined with chemotherapy plus Toripalimab or not for the first-line treatment of SCLC, and maintenance therapy are Surufatinib combined with Toripalimab or not.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and voluntarily sign informed consent;
2. Age: ≥18 years old;
3. Expected survival period ≥ 3 months;
4. Adavanced small cell lung cancer confirmed by histology ;
5. According to the RECIST 1.1 standard, the patient has at least one target lesion with a measurable diameter;
6. ECOG PS: 0-1;
7. Laboratory test indicators must meet the following requirements: Hematology: white blood cells ≥4.0×10^9/L, neutrophils ≥2.0×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥90g/L. Liver function: serum bilirubin is lower than 1.5 times the maximum normal value; for patients without liver metastasis: ALT and AST are lower than 2.5 times the maximum normal value; for patients with liver metastasis: ALT and AST are lower than 5 times the maximum normal value ; Measured or calculated creatinine clearance: According to the Cockcroft-Gault formula (using actual body weight), patients receiving cisplatin treatment>60mL/min, and patients receiving carboplatin treatment>45mL/min;
8. Good compliance and follow-up;
9. The urine or serum pregnancy test results of premenopausal women were negative.

Exclusion Criteria:

1. Patients with symptomatic brain metastases;
2. People with hypertension who cannot be well controlled by double antihypertensive drug (systolic blood pressure≥140 mmHg, diastolic blood pressure≥90 mmHg);
3. Urine routine test showed urine protein ≥+++ and confirmed 24-hour urine protein quantification>3.0g;

5.Cardiovascular disease history: congestive heart failure> New York Heart Association (NYHA) standard II, patients with active coronary artery disease (those with myocardial infarction 6 months before enrollment can be enrolled), arrhythmia requiring treatment (Allows to take beta blockers or digoxin); 6.Active severe clinical infections (>NCI-CTCAE 5.0 version 2 infection criteria), including tuberculosis (clinical evaluation, including clinical history, physical examination, imaging findings and TB examination in line with local clinical practice), hepatitis B (known HBV Surface antigen [HbsAg] positive), hepatitis C or human immunodeficiency virus (HIV 1/2 antibody positive). Patients who have previously had HBV infection or have been cured (defined as the presence of hepatitis B core IgG antibodies and the absence of HBsAg) are eligible. Hepatitis C virus (HCV) antibody-positive patients are only eligible if the HCV RNA polymerase chain reaction is negative; 7.Patients with bleeding tendency or coagulation disorders, (14 days before randomization must meet: INR is within the normal range without the use of anticoagulants); 8.In the past 2 years, there are active autoimmune diseases that require systemic treatment (such as corticosteroids or immunosuppressive drugs), and related alternative treatments (such as thyroxine, insulin, or physiological corticosteroid replacement for renal or pituitary insufficiency) are allowed treatment); 9.Those who have received live vaccination within 4 weeks before the start of treatment; 10.Those who had suffered from tumors other than small cell lung cancer within 5 years before being enrolled in this study. Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor; 11.Severe unhealed wounds, ulcers or fractures; 12.Patients who are pregnant or breastfeeding ; 13.Any unstable conditions may endanger the safety of patients and affect their compliance with research; 14.Researchers think it is inappropriate to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival(PFS) | up to 24 months

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 24 months
Overall Survival(OS) | up to 24 months
Disease control rate(DCR) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Y, Huang Y, Yang Y, Zhao Y, Zhou T, Chen G, Zhao S, Zhou H, Ma Y, Hong S, Zhao H, Zhang L, Fang W. Surufatinib plus toripalimab combined with etoposide and cisplatin as first-line treatment in advanced small-cell lung cancer patients: a phase Ib/II trial. Signal Transduct Target Ther. 2024 Sep 27;9(1):255. doi: 10.1038/s41392-024-01974-2. PMID 39327433